CLINICAL TRIAL: NCT01931969
Title: Comparison of Internal Jugular Vein Catheterization Entry Points Determined by Ultrasonography Versus the Central Landmark Guided Method
Brief Title: Central Landmark vs USG for IJV Catheterization
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ozlem Can, MD, Instructor in Department of Anesthesiology And Intensive Care, Ankara University
Other Study IDs: CLM vs USG for RIJVC; CLMUSGRIJVC (Registry Identifier: Ankara University)
Record Dates: First submitted 2013-08-22; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Value of Central Landmark Method for Juguler Vein Catheterization
Keywords: Vein catheterization; Ultrasound; Landmark; Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IJVC intervention

SUMMARY:
This study is planned to compare right internal jugular vein catheterization entry points determined by ultrasound and the central landmark guided method, and the relationship of each with sternocleidomastoid muscle length and body mass index.

ELIGIBILITY:
Inclusion Criteria:

-patients undergoing cardiovascular surgery who needed to have internal jugular vein catheterization aged 18y or older-

Exclusion Criteria:

-previous neck surgery, burns, limited neck movement, diffuse goiter or bleeding problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing cardiovascular surgery who needed to have internal jugular vein catheterization
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Success rate with the Central Landmark Method | 1 mounth

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Ankara, Turkey (Türkiye)